CLINICAL TRIAL: NCT07367698
Title: Clinical Investigation Evaluating Medical Grade Polycaprolactone (PCL) Breast Scaffold Implantation in Conjunction With Autologous Fat Grafting for Breast Implant Revision Surgery
Brief Title: Scaffold-guided Breast Implant Revision Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: BellaSeno Pty Ltd (Industry)
Responsible Party: Sponsor
Organization: BellaSeno GmbH (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2025-BRV-005
Record Dates: First submitted 2026-01-09; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Breast Implant Revision; Breast Augmentation Complications
Keywords: Breast scaffold; PCL Scaffold; Absorbable Implant; Regenerative Medicine; Implant Removal; Breast Surgery; Clinical Safety and Performance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Implantation of the PCL Breast scaffold with autologous fat grafting (Experimental): Implantation of the PCL Breast Scaffold with autologous fat graft for breast augmentation implant revision
  Interventions: Device: Implantation of the PCL Breast scaffold with autologous fat grafting

INTERVENTIONS:
Device: Implantation of the PCL Breast scaffold with autologous fat grafting — The PCL Breast Scaffold is implanted either immediately following the removal of a silicone implant or during a delayed procedure. The surgery uses the same surgical pocket from the previous augmentation for insertion of the PCL Breast Scaffold, or, if implants have been previously removed, a new surgical pocket will be created. The PI will ensure accurate placement and secure fixation of the scaffold in the desired anatomical position. Autologous fat grafting (AFG) is then performed: the fat cells are harvested from the abdomen and/or thighs and injected into the implanted scaffold at the time of initial implantation. Lastly, after the AFG has been performed, wound closure and dressing will be conducted as per standard procedure. Sterile bandaging shall be initially applied and the wound reviewed daily whilst an inpatient.
  In conjunction with scaffold implantation, concurrent breast procedures may be performed on a case-by-case basis (e.g., Mastopexy,...).

SUMMARY:
The objective of this clinical trial is to generate robust data that demonstrates clinical performance and safety of a polycaprolactone (PCL) breast scaffold combined with autologous fat grafting (AFG) in women who seek a revision surgery of a breast implant used for breast augmentation. The material (PCL) has been in clinical use for many decades and is absorbable. This study follows the successful completion of a 2-year evaluation of the safety and feasibility of this technique performed by the Royal Brisbane and Women's Hospital (ClinicalTrials.gov ID: NCT05437757).

The main question it aims to answer is: "Is PCL Breast Scaffold with autologous fat graft a safe and effective method of soft tissue reconstruction following breast implant revision?".

Participants will:

* Undergo removal of their existing silicone breast implant (if not previously removed),
* Receive implantation of a PCL Breast Scaffold combined with autologous fat grafting (AFG), and
* Attend follow-up visits at 1 week, 3 months, 6 months, and annually for up to 5 years for clinical assessments and questionnaires.

ELIGIBILITY:
Inclusion Criteria

To be eligible to participate in this clinical investigation, patients must meet ALL of the following criteria:

1. Genetically female
2. Patients, age from 18 years old undergoing surgical revision of bilateral breast implants originally placed for cosmetic augmentation
3. Patients with a target volume that can be treated with the available catalogue of PCL scaffold sizes
4. Eligible to undergo MRI (i.e., no implanted incompatible metal or metal devices, no history of severe claustrophobia)
5. Agree to maintain their weight (i.e., within 5%) by not making any major changes in diet or lifestyle during the study
6. Agree to not undergo any elective cosmetic surgery on her breasts for a minimum of 3 years following implantation of the investigational device

Exclusion Criteria

Patients may not participate in the clinical investigation if they meet ANY of the following criteria:

1. Based on the judgement of the Investigator, inadequate sites/ volume for harvesting the fat graft
2. Medical history of any malignant condition in the breast or chest wall region
3. Medical history of BRCA 1 or BRCA 2 Mutation
4. Abnormal findings on diagnostic imaging in the breast(s) intended for treatment within one year of study enrolment
5. Prior history of infection in the breast in the preceding 12 months
6. Prior surgery involving the breast in the preceding 12 months (except any previous removal of silicone implant)
7. Breast feeding in the preceding 12 months
8. Any local infection or rash within or close to the surgical fields (harvest site(s) or breasts)
9. Medical history of Breast Implant-Associated Anaplastic Large Cell Lymphoma (BIA ALCL) or Breast Implant Associated Squamous Cell Carcinoma (BIA-SCC)
10. The patient has any disease, that is clinically known to impact wound healing ability
11. Known history of immunodeficiency including HIV, concomitant systemic corticosteroid therapy, chemotherapy, synchronous haematological malignancy or other cause for secondary/primary immunodeficiency
12. Micro or macro angiopathia
13. Uncontrolled endocrine disorders
14. Clotting disorders, including thromboembolism
15. Known severe concurrent or intercurrent illness including cardiovascular, respiratory or immunological illness, psychiatric disorders, alcohol or chemical dependence, possible allergies that would, in the opinion of the Investigator, compromise safety or compliance, or interfere with interpretation of study results
16. Polycaprolactone (PCL) allergy
17. Currently pregnant or breast feeding, or who are planning to become pregnant within 5 years after the breast surgery
18. Actively smoking or have a history of smoking (patient with a history of smoking may still be eligible pending assessment by investigating team and documentation of rationale)
19. Actively using recreational drugs or have a history of use of recreational drugs (patients with a history of use of recreational drugs may still be eligible pending assessment by investigating team and documentation of rationale)
20. Known allergies to MRI contrast agents
21. Unable or unwilling to comply with the treatment protocol
22. Unwilling or unable to provide fully informed consent including but not limited to patients with intellectual or mental impairment
23. Currently enrolled or has plans to enrol in another clinical study that would interfere with this study, unless it is retrospective or observational
24. Any patient condition that, in the Investigator's opinion, would preclude the use of the study device, interfere with the evaluation of the device or breast related outcomes, or would preclude participation in the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Females
Enrollment: 73 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2032-01 (Estimated); Study Completion 2032-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the occurrence rate of moderate and severe device-related (probable and causal) AEs aftersurgical revision of permanent breast implants within 12 months | Assessed at post-surgery, at 1 week and at 3-, 6- and 12-month post sugery
  Number of moderate and severe AEs with a probable or causal relationship to the device falling under pre-defined category over time

SECONDARY OUTCOMES:
Breast revision surgery rate | Assessed at post-surgery and at 1-week, 3-month, 6-month, 1-year, 2-year, 3-year, 4-year and 5-year post-surgery
  Number of breast revision surgeries categorized by reason and time
Rate and severity of all AEs related to device and/or procedure | Assessed at post-surgery, 1-week, 3-month, 6-month, 1-year, 2-year, 3-year, 4-year and 5-year post-surgery
  Number of AEs categorised by relationship with device and/or procedure (possible, probable, causal), severity and type over time
Total breast volume retention (3D Imaging) | Assessed at enrolment and at 3-month, 6-month, 1-year, 2-year, 3-year, 5-year post-surgery
  Total breast volume primarily assessed through 3D imaging. Supportive data generated by:
  * Dynamic contrast enhanced Magnetic Resonance Imaging (DCE-MRI);
  * Breast anthropomorphic measurements taken with tape measure or with Vectra imaging system (Sternal notch to nipple (SN-N), Nipple to Inframammary Fold (N-IMF), Overbust measurement, Underbust measurement, Chest circumference at highest projection);
  * Digital photos
Assessment of patient satisfaction, quality of life, body image, and psychological well-being using validated questionnaires (BREAST-Q) | Assessed at enrolment and at 3-month, 6-month, 1-year, 2-year, 3-year, 4-year, 5-year post-surgery
  Patient-reported outcomes will be measured using the validated BREAST-Q questionnaire. Results are reported as a transformed score range from 0 to 100, with higher scores reflecting a better outcome.
Assessment of patient satisfaction, quality of life, body image, and psychological well-being using a 5-point Likert scale questionnaire | Assessed at 3-month, 6-month, 1-year, 2-year, 3-year, 4-year, 5-year post-surgery
  Patient-reported outcomes will be measured through a 5-point Likert scale questionnaire. Scores range from 1 to 5, with higher scores indicating better outcomes.
Assessment of surgical usability and surgeon satisfaction using a 5-point Likert scale questionnaire | Assessed at surgery and at 3-month, 6-month, 1-year, 2-year, 3-year, 4-year, 5-year post-surgery
  The 5-point Likert scale questionnaire is administered to the PIs performing the surgical procedure. Scores range from 1 to 5, with higher scores indicating a better usability and greater surgeon satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Professor Owen Ung, Principal Investigator — Royal Brisbane and Women's Hospital, Herston Biofabrication Institute
Locations (6):
- Australia (3):
  - Macquarie University Hospital, Sydney, New South Wales
  - Westmead Hospital, Lakeview Private Hospital, Sydney, New South Wales
  - Royal Brisbane and Women's Hospital (RBWH), Herston Biofabrication Institute (HBI), Brisbane, Queensland
- Zealand University Hospital, Roskilde, Region Sjælland, Denmark
- Germany (2):
  - Evangelisches Krankenhaus Göttingen-Weende, Göttingen, Lower Saxony
  - Universitätsklinikum Münster, Münster, North Rhine-Westphalia

IPD SHARING:
Plan to Share IPD: No